CLINICAL TRIAL: NCT00430157
Title: An 8 Day, Randomised, Double Blinded, Placebo-controlled 2-way Crossover Trial of Repeat Doses of Intranasal GSK256066 and Placebo in the Vienna Challenge Chamber in Subjects With Seasonal Allergic Rhinitis (SAR)
Brief Title: Trial With Allergic Rhinitis Patients Taking GSK256066 Versus Placebo In A Pollen Challenge Chamber
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IPR107498
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Rhinitis, Allergic, Seasonal; Seasonal Allergic Rhinitis
Keywords: Vienna Challenge Chamber; Seasonal Allergic Rhinitis; Inflammation
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Inflammation | interventions — 6-((3-((dimethylamino)carbonyl)phenyl)sulfonyl)-8-methyl-4-((3-methyloxyphenyl)amino)-3-quinolinecarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK256066

SUMMARY:
This study is in patients with seasonal allergic rhinitis (SAR) and will compare the effect versus placebo of repeat doses of intranasal GSK256066 using the Vienna Challenge Chamber. GSK256066 is a potent and highly selective phosphodiesterase-4 (PDE4) inhibitor, currently in development by GSK for the treatment of allergic rhinitis, asthma and COPD.

Subjects will be selected on the basis that they display a defined moderate response to the pre-determined dose used.

This study aims to explore the actions of repeat doses of intranasal GSK256066 in patients with Seasonal Allergic Rhinitis in the Vienna Challenge Chamber compared to placebo.

12-lead ECG, vital signs and adverse event enquiries will be made throughout the study. Nasal examination, symptom scores (TNSS), nasal lavage, nasal scrape and allergen challenge assessments will also be performed at various time points throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* The subject is healthy.
* They are aged 18 to 50 years inclusive.
* Body mass index less than 29.0 kg/m² with weight range of 55.0kg (females 50kg) to 95.0kg inclusive.
* They have a history of seasonal allergic rhinitis
* They exhibit a moderate response to 1500 grass pollen grains/m3 after 2h in the Vienna Challenge Chamber,
* They have a positive skin prick test for grass pollen at or within the 12 months preceding the screening visit.
* They have a positive RAST for grass pollen at or within the 12 months preceding the screening visit.
* They are current non-smokers who have not used any tobacco products in the 6 months preceding the screening visit
* They must have a baseline FEV1>80% predicted and a baseline FEV1 (maximum recorded value)/ FVC (associated value)>70% predicted.

Exclusion Criteria:

* Pregnant or nursing females.
* Women of childbearing potential who are unwilling or unable to use an appropriate method of contraception.
* any structural nasal abnormalities or nasal polyposis, a history of frequent nosebleeds, recent nasal surgery or recent (within 2 weeks) or ongoing upper respiratory tract infection.
* The subject is likely to be unable to abstain from salbutamol use for 8 hours before a challenge
* The subject has a history of drug or other allergy
* The subject is concurrently participating in another clinical study in the past 3 months
* A supine blood pressure that is persistently higher than 140/90 millimetres of mercury (mmHg) at screening
* A supine mean heart rate outside the range 40-90 beats per minute (bpm) at screening.
* The subject has donated a unit of blood within the previous 3 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2007-01

PRIMARY OUTCOMES:
Weighted mean total nasal symptom score (TNSS) (sneeze, itch, rhinorrhoea and obstruction) | 1-4h post-dose period spent in the Vienna Challenge Chamber on Day 7

SECONDARY OUTCOMES:
Weighted mean total nasal symptom score (TNSS) (sneeze, itch, rhinorrhoea and obstruction) | 1-4h post morning dose period spent in the Vienna Challenge Chamber on Day 2.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Vienna, Austria